CLINICAL TRIAL: NCT02637297
Title: Hypnosis for Pain Management With Cancer Survivors
Brief Title: Hypnotherapy in Treating Chronic Pain in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH); American Nurses Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9445; NCI-2015-01868 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9445 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH); T32NR013456 (NIH)
Record Dates: First submitted 2015-12-04; First posted 2015-12-22 (Estimated); Last update posted 2017-08-21 (Actual); Status verified 2017-08

CONDITIONS: Anxiety; Cancer Survivor; Chronic Pain; Depression; Sleep Disorder
MeSH Terms: conditions — Anxiety Disorders; Chronic Pain; Depression; Sleep Wake Disorders | interventions — Hypnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group I (immediate intervention group) (Experimental): Participants undergo hypnotherapy session over 20-30 minutes using a standardized script for pain reduction that contains post-hypnotic suggestions for permanence of hypnotherapy benefits. The hypnotherapy session is recorded and the participant listens to the recording daily for 4 weeks.
  Interventions: Procedure: Hypnotherapy; Other: Questionnaire Administration
- Group II (wait-list control group) (Active Comparator): At week 5, participants undergo hypnotherapy session over 20-30 minutes using a standardized script for pain reduction that contains post-hypnotic suggestions for permanence of hypnotherapy benefits. The hypnotherapy session is recorded and the participant listens to the recording daily for 4 weeks.
  Interventions: Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Hypnotherapy — Undergo hypnotherapy
  Other Names: Hypnosis
  Arms: Group I (immediate intervention group)
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This randomized pilot clinical trial studies hypnotherapy in treating chronic pain in cancer survivors. Hypnotherapy is a state of concentration and focused attention which can provide more control over the experience of acute and chronic pain and its impact and may provide comfort, maximize function, and improve quality of life in cancer survivors.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the feasibility (recruitment, attrition, adherence, logistical issues) of delivering the hypnosis (hypnotherapy) intervention to cancer survivors with chronic pain.

II. To evaluate the acceptability of the hypnosis intervention among cancer survivors with chronic pain.

III. To explore preliminary efficacy (estimate effect size) of hypnosis in relieving pain and improving associated anxiety and functional performance at 4 weeks and 8 weeks compared to a wait-list control.

OUTLINE: Participants are randomized to 1 of 2 groups.

IMMEDIATE INTERVENTION GROUP: Participants undergo hypnotherapy session over 20-30 minutes using a standardized script for pain reduction that contains post-hypnotic suggestions for permanence of hypnotherapy benefits. The hypnotherapy session is recorded and the participant listens to the recording daily for 4 weeks.

WAIT-LIST CONTROL GROUP: At week 5, participants undergo hypnotherapy session over 20-30 minutes using a standardized script for pain reduction that contains post-hypnotic suggestions for permanence of hypnotherapy benefits. The hypnotherapy session is recorded and the participant listens to the recording daily for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Self-report of moderate or higher pain on average during the last week (> 3 on a 0-10 pain intensity numeric scale)
* Completed active cancer treatment other than maintenance therapy >= 3 months ago
* Functional fluency in English
* Mentally and physically able to participate and complete surveys over the phone

Exclusion Criteria:

* Chronic pain is not cancer-related

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-01-08 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2017-08-03 (Actual)

PRIMARY OUTCOMES:
Acceptability of hypnotherapy determined by structured phone interviews with participants | At week 8
  Transcribed interview data and open-ended responses from the pre- post-Intervention Questionnaire will be organized in ATLAS.ti. Content analysis will be used to understand the hypnosis experience. Consensus on key ideas and concepts will be obtained by the Lead Sub-Investigator and research assistant after reading and coding each transcript separately.
Change in beliefs on how well the treatment might work, as measured by the Credibility/Expectancy Questionnaire | Baseline to up to 8 weeks
  To evaluate the effects of the intervention on efficacy endpoints, general linear modeling will be used. Participants will be a random effect. There will be 2 fixed effects (time, group) and 1 interaction effect (time X group). The interaction between group x time will show if the groups change differentially (whether intervention moderates change in outcome). Within the wait-list, O2 and O3 will be compared (paired t-test) to see if the wait-list replicates the immediate group's results. Within the immediate group, sustained effects of post-intervention results will be assessed by testing for
Change in imaginative involvement as measured by the Tellegen Absorption Scale | Baseline to up to 8 weeks
  To evaluate the effects of the intervention on efficacy endpoints, general linear modeling will be used. Participants will be a random effect. There will be 2 fixed effects (time, group) and 1 interaction effect (time X group). The interaction between group x time will show if the groups change differentially (whether intervention moderates change in outcome). Within the wait-list, O2 and O3 will be compared (paired t-test) to see if the wait-list replicates the immediate group's results. Within the immediate group, sustained effects of post-intervention results will be assessed by testing for
Change in pain and anxiety, as measured using the patient diary | Baseline to up to 8 weeks
  To evaluate the effects of the intervention on efficacy endpoints, general linear modeling will be used. Participants will be a random effect. There will be 2 fixed effects (time, group) and 1 interaction effect (time X group). The interaction between group x time will show if the groups change differentially (whether intervention moderates change in outcome). Within the wait-list, O2 and O3 will be compared (paired t-test) to see if the wait-list replicates the immediate group's results. Within the immediate group, sustained effects of post-intervention results will be assessed by testing for
Change in pain and anxiety, as measured using the Pre- Post-Intervention Questionnaire | Baseline to up to 8 weeks
  To evaluate the effects of the intervention on efficacy endpoints, general linear modeling will be used. Participants will be a random effect. There will be 2 fixed effects (time, group) and 1 interaction effect (time X group). The interaction between group x time will show if the groups change differentially (whether intervention moderates change in outcome). Within the wait-list, O2 and O3 will be compared (paired t-test) to see if the wait-list replicates the immediate group's results. Within the immediate group, sustained effects of post-intervention results will be assessed by testing for
Change in pain-associated anxiety, measured using the Pain Catastrophizing Scale | Up to 8 weeks
  To evaluate effects of intervention on efficacy endpoints, general linear modeling will be used. Participants will be a random effect. There will be 2 fixed effects (time and group) & 1 interaction effect (time X group). Interaction between group x time will tell if groups change differentially (whether intervention moderates change in outcome). Within wait-list, O2 & O3 will be compared (paired t-test) to see if wait-list replicates immediate group's results. Within immediate group, sustained effects of post-intervention results will be assessed by testing for change across time to O3. During
Change in Patient Reported Outcomes Measurement Information System-29 scores (measures function, anxiety, depression, fatigue, sleep, and pain interference and intensity) | Baseline to up to 8 weeks
  To evaluate the effects of the intervention on efficacy endpoints, general linear modeling will be used. Participants will be a random effect. There will be 2 fixed effects (time, group) and 1 interaction effect (time X group). The interaction between group x time will show if the groups change differentially (whether intervention moderates change in outcome). Within the wait-list, O2 and O3 will be compared (paired t-test) to see if the wait-list replicates the immediate group's results. Within the immediate group, sustained effects of post-intervention results will be assessed by testing for
Feasibility of delivering hypnotherapy in terms of recruitment, attrition, adherence, and logistical issues | Up to 12 months
  A Consort flow diagram will be maintained to record the number of patients who were invited to participate in the study, number of patients who declined to participate and reasons why, number of patients who did not complete the study and reasons why, and adherence to using the intervention. Descriptive statistics (frequency counts, percentages) will be used to analyze the study recruitment, enrollment, and attrition data.
Patient demographics, as measured by the Demographic Questionnaire | Baseline
  Demographic variables will be analyzed using descriptive and inferential statistics. In order to examine variability and estimate effect sizes, the analysis needed in a larger trial will be modeled. Baseline demographic and dependent variables for the immediate and wait-list condition groups will be compared with Chi-square or independent t-tests.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Shannon Dorcy, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States